CLINICAL TRIAL: NCT03475251
Title: A Phase Ia/Ib, Open-Label, Multiple-Dose, Dose-Escalation and Expansion Study of the Anti-PD-1 Monoclonal Antibody CS1003 in Subjects With Advanced Solid Tumors
Brief Title: A Study of CS1003 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1003-101; ACTRN12618000382279 (Registry Identifier: The Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — CS-1003; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CS1003 (Experimental)
  Interventions: Biological: CS1003
- CS1003 + regorafenib (Experimental)
  Interventions: Biological: CS1003; Drug: Regorafenib

INTERVENTIONS:
Biological: CS1003 — In the dose escalation part, the dose levels will be escalated following a modified 3+3 dose escalation scheme. In the dose expansion part, patients will be assigned to different groups based on their tumor type.
  Arms: CS1003
Biological: CS1003 — CS1003 to be intravenously administered at the dose level determined during the dose escalation part
  Arms: CS1003 + regorafenib
Drug: Regorafenib — Regorafenib to be orally administered at the protocol-specified dose level, once daily for the first 21 days of each 28-day cycle
  Arms: CS1003 + regorafenib

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetic profile and treatment effect of a new drug known as CS1003 in patients with advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed advanced or metastatic solid tumor and have progressed, are intolerant to, refuse to accept or do not have access to standard therapy.
2. ECOG performance status of 0 or 1.
3. Subjects with evaluable but non-measurable lesion are eligible for Phase Ia. Subjects must have at least one measurable lesion per RECIST Version 1.1 to be eligible for Phase Ib.
4. Archived tumor tissue samples need to be collected, or subjects consent to undergo pre-treatment biopsy if archived sample is not available.
5. Life expectancy ≥ 3 months.
6. Subject must have adequate organ function.
7. Use of effective contraception (males and females).

Exclusion Criteria:

1. Subjects with known symptomatic or untreated brain metastasis or other CNS metastasis.
2. Subjects with active autoimmune diseases or history of autoimmune diseases.
3. Subjects who have to receive glucocorticoids (prednisone at > 10 mg/day or equivalent) or other immunosuppression within 14 days prior to the first dose of CS1003.
4. Subjects with other malignant tumor(s) in the past 2 years are not eligible for Phase Ib, except for those with basal cell carcinoma, in situ breast cancer and cervical carcinoma in situ who have undergone radical treatment.
5. Subjects who have received any immune checkpoint treatment, including PD-1, PD-L1, etc.
6. Receipt of chemotherapy, targeted therapy, or any other anti-cancer systemic treatment within 2 weeks prior to the first dose of CS1003.
7. Receipt of major surgical procedure or wide field of radiation within 28 days prior to the first dose of CS1003, local radiotherapy within 14 days prior to the first dose of CS1003, or radioactive agents within 56 days before the first dose of CS1003.
8. Receipt of Chinese herbal medicine or Chinese prepared medicine within 7 days prior to the first dose of CS1003.
9. Receipt of live vaccine within 28 days prior to the first dose of CS1003.
10. History of interstitial lung disease or non-infectious pneumonitis, except for those induced by radiation therapies.
11. History of HIV infection.
12. Subjects with active Hepatitis B and C infection (HBV DNA ≥ 1000 cps/mL or 200 IU/mL) requiring therapy.
13. Subjects with active infection of tuberculosis.
14. Subjects with signs or symptoms of any active infection requiring systemic therapy.
15. History of organ transplantation.
16. Unresolved toxicities from prior anti-cancer therapy.
17. History of any irAE of Grade ≥ 3.
18. History of uncontrolled allergic asthma and serious hypersensitive reaction to monoclonal antibodies.
19. History of alcoholism or drugs abuse.
20. Subjects with major cardiovascular diseases.
21. Any condition that, in the opinion of the investigator or sponsor, would jeopardize compliance.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From the day of first dose to 30 days after last dose of CS1003

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | From the day of first dose to 30 days after last dose of CS1003
Maximum plasma concentration (Cmax) | From the day of first dose to 30 days after last dose of CS1003
Time to reach maximum plasma concentration (Tmax) | From the day of first dose to 30 days after last dose of CS1003
Terminal elimination half-life (t1/2) | From the day of first dose to 30 days after last dose of CS1003
Disease assessment by CT/MRI scan | To be performed every 9 weeks during treatment period (up to 2 years) and within 30 days after last dose of CS1003
Anti-CS1003 antibody | From the day of first dose to 30 days after last dose of CS1003

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia

REFERENCES:
- [Derived] Gong J, Guo Y, Zhang Y, Ba Y, Chen T, Li W, Zhou C, Wang M, Yang H, Zhou Y, Cai Q, Wang Z, Huang G, Zhang W, Su R, Cai Z, Yue Z, Dou J, Li P, Wu R, Tse AN, Shen L. A Phase 1a/1b Dose Escalation/Expansion Study of the Anti-PD-1 Monoclonal Antibody Nofazinlimab in Chinese Patients with Solid Tumors or Lymphoma. Target Oncol. 2024 Sep;19(5):723-733. doi: 10.1007/s11523-024-01091-8. Epub 2024 Sep 4. PMID 39231855
- [Derived] Day D, Park JJ, Coward J, Markman B, Lemech C, Kuo JC, Prawira A, Brown MP, Bishnoi S, Kotasek D, Strother RM, Cosman R, Su R, Ma Y, Yue Z, Hu HH, Wu R, Li P, Tse AN. A first-in-human phase 1 study of nofazinlimab, an anti-PD-1 antibody, in advanced solid tumors and in combination with regorafenib in metastatic colorectal cancer. Br J Cancer. 2023 Nov;129(10):1608-1618. doi: 10.1038/s41416-023-02431-7. Epub 2023 Sep 20. PMID 37731023